CLINICAL TRIAL: NCT00533026
Title: Evaluation of the Effect of Duloxetine on the Pharmacodynamics of Warfarin at Steady-State in Healthy Subjects
Brief Title: Duloxetine - Warfarin Pharmacodynamic Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 11707; F1J-MC-HMFP
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Last update posted 2008-10-02 (Estimated); Status verified 2008-09

CONDITIONS: Anticoagulant Effect of Warfarin When Taken With Duloxetine.
MeSH Terms: interventions — Duloxetine Hydrochloride; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Subjects received warfarin QD, PO for approximately 12 days. Subjects with stabilized INR after approximately 12 days continued to receive warfarin QD, PO for an additional 14 days and also received duloxetine 60mg QD, PO for the 14 days. Duloxetine doses were tapered, subjects received 30mg QD, PO for 4 days. No warfarin was received during the taper phase.
  Interventions: Drug: Duloxetine; Drug: Warfarin
- B (Active Comparator): Subjects received warfarin QD, PO for approximately 12 days. Subjects with stabilized INR after approximately 12 days continued to receive warfarin QD, PO for an additional 14 days and also received duloxetine 60 mg QD, PO for 4 days followed by duloxetine 120 mg QD, PO for 10 days. Duloxetine doses were tapered, subjects received 60mg QD, PO for 4 days followed by 30mg QD, PO for 4 days. No warfarin was received during the taper phase.
  Interventions: Drug: Duloxetine; Drug: Warfarin

INTERVENTIONS:
Drug: Duloxetine
  Other Names: LY248686; Cymbalta
Drug: Warfarin

SUMMARY:
To evaluate the blood clotting effects of multiple doses of warfarin at steady state when taken at the same time as multiple doses of duloxetine as measured by changes in the International Normalised Ratio. All subjects will begin dosing with warfarin, then after approximately 12 days, duloxetine 60 mg is added and subjects with stabilized INR will either continue dosing at 60 mg or have a dose increase to 120 mg.

ELIGIBILITY:
Inclusion Criteria:

Healthy men or women between ages 18 and 64 years.

Exclusion Criteria:

Have a personal history, family history of, or current evidence of: a bleeding disorder, have Positive Faecal Occult Blood (FOB) sample at screening, significant neuropsychiatric disease (including a history of suicide attempts or who have exhibited suicidal ideation or who are at significant risk to commit suicide, as judged by the investigator), significant active respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders.

Use or intended use of aspirin or NSAIDs within 2 weeks prior to first dosing.

Subjects who have an average weekly alcohol intake that exceeds 28 units per week (males) and 21 units per week (females). Subjects who smoke more than 5 cigarettes per day.

Use or intended us of a drug that inhibits or induces CYP1A2 or inhibits CYP2D6 within 2 weeks prior to first dosing occasion or during the study.

Have received any drug that acts as a monoamine oxidase inhibitor (MAOI) within 2 weeks prior to first dosing occasion or have a potential need to use an MAOI during the conduct of this study or within 2 weeks after discontinuation of study drug.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2007-07; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
International Normalized Ratio (INR) | 58 days

SECONDARY OUTCOMES:
Effect of duloxetine on pharmacokinetics of warfarin. | 58 days
Safety/ tolerability of duloxetine and warfarin given in combination. | 58 days
Bleeding times when duloxetine and warfarin are given in combination. | 58 days

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559), Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Leeds, West Yorkshire, United Kingdom

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com